CLINICAL TRIAL: NCT02536456
Title: China PEACE Million Persons Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20150823
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Disease
Keywords: screening; counseling; follow-up; cardiovascular disease; population-based project; China
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For each high-risk subject, a 6mL whole blood sample is collected in an EDTA vacuum tube.A 10mL urine sample is also collected.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
China PEACE Millions Persons Project is a national screening project for cardiovascular disease in China. This Project was approved by National Health and Family Planning Commission (NHFPC), China and founded by Ministry of Finance, China in 2014.

The specific objectives of the project are to:

1. identify subjects at high-risk of CVD and provide counseling for medication and lifestyle improvements
2. evaluate the feasibility of such screening methods for subjects at high risk of CVD, and to assess the effect of health counseling on CVD incidence rates and risk factors control
3. inform future intervention and long-term follow up efforts for primary and secondary CVD prevention in China.

ELIGIBILITY:
Inclusion Criteria:

1. 35 - 75 years old
2. registered in the Hukou of the selected region
3. sign the consent form

Exclusion Criteria:

-

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents from the communities or villages in selected sites
Sampling Method: Non-Probability Sample
Enrollment: 4000000 (Estimated)
Dates: Start 2014-07; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Cardiovascular diseases | 5 years
  Number of new cardiovascular diseases in high-risk subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu X, Lin S, Zhang H, Zhang X, Wu C, Chen B, Yang Y, Cui J, Xu W, Song L, Yang H, He W, Zhang Y, Li X, Lu J. Association of HDL subclass components with all-cause and cardiovascular mortality: a prospective cohort study based on the ChinaHEART project. Lipids Health Dis. 2026 Jan 27. doi: 10.1186/s12944-026-02874-w. Online ahead of print. PMID 41593465
- [Derived] Wang Y, Peng K, Xu W, Huang X, Liu X, Li Y, Lu J, Yang Y, Chen B, Shi Y, Han G, Zhang X, Cui J, Song L, Tian A, Runsi W, Wang C, Tian Y, Wu Y, Lin C, Peng W, Li X, Hu S. Cardiovascular disease-specific and all-cause mortality across socioeconomic status and lifestyles among patients with established cardiovascular disease in communities of China: data from a national population-based cohort. Heart. 2025 Oct 29;111(22):1092-1100. doi: 10.1136/heartjnl-2024-324766. PMID 40081938
- [Derived] Wang R, Wang Y, Lu J, Li Y, Wu C, Yang Y, Cui J, Xu W, Song L, Yang H, He W, Zhang Y, Zhang X, Li X, Hu S. Forecasting cardiovascular disease risk and burden in China from 2020 to 2030: a simulation study based on a nationwide cohort. Heart. 2025 Feb 12;111(5):205-211. doi: 10.1136/heartjnl-2024-324650. PMID 39638429
- [Derived] China PEACE Collaborative Group; Zhou T, Wang Y, Zhang H, Wu C, Tian N, Cui J, Bai X, Yang Y, Zhang X, Lu Y, Spatz ES, Ross JS, Krumholz HM, Lu J, Li X, Hu S. Primary care institutional characteristics associated with hypertension awareness, treatment, and control in the China PEACE-Million Persons Project and primary health-care survey: a cross-sectional study. Lancet Glob Health. 2023 Jan;11(1):e83-e94. doi: 10.1016/S2214-109X(22)00428-4. PMID 36521957
- [Derived] Lu J, Xuan S, Downing NS, Wu C, Li L, Krumholz HM, Jiang L. Protocol for the China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Million Persons Project pilot. BMJ Open. 2016 Jan 4;6(1):e010200. doi: 10.1136/bmjopen-2015-010200. PMID 26729395